CLINICAL TRIAL: NCT03709394
Title: Two Different Techniques for Ultrasound Guided Peripheral Venous Catheter Insertion in Pre-hospital Emergency Care - Randomized Study
Brief Title: Pre-hospital Ultrasound Guided Peripheral Venous Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Head physician for science and research, Emergency Medical Service of the Central Bohemian Region, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01
Record Dates: First submitted 2018-05-08; First posted 2018-10-17 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Prehospital
Keywords: ultrasound; peripheral venous catheter

STUDY DESIGN:
Intervention Model Description: Prospective randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Full utrasound guidance (Active Comparator): Full utrasound guidance of cathether insertion. Intervention: Ultrasound portable device used for the identification of the target vein and for the ultrasound control of proper catheter placement during the procedure of peripheral venous cannula insertion.
  Interventions: Procedure: Full utrasound guidance
- Group B: Partial ultrasound guidance (Active Comparator): Catheter insertion under partial ultrasound guidance. Intervention: Ultrasound portable device used only for the identification of the target vein, the catheter placement will be done by conventional approach.
  Interventions: Procedure: Partial ultrasound guidance
- Group C: No ultrasound guidance (Active Comparator): Catheter insertion by conventional approach, without ultrasound guidance
  Interventions: Procedure: No ultrasound guidance

INTERVENTIONS:
Procedure: Full utrasound guidance — The target vein is directly identified by portable ultrasound device and the complete procedure of peripheral venous cathether insertion is controlled by ultrasound guidance in real time
  Arms: Group A: Full utrasound guidance
Procedure: Partial ultrasound guidance — The target vein is directly identified by ultrasound but the procedure of peripheral venous cathether insertion is performed conventionally, without ultrasound guidance
  Arms: Group B: Partial ultrasound guidance
Procedure: No ultrasound guidance — The target vein is identified and peripheral venous catheter is inserted by conventional approach without use of any guiding devices
  Arms: Group C: No ultrasound guidance

SUMMARY:
This study evaluates two different techniques for ultrasound guided peripheral venous catheter insertion in pre-hospital emergency care in comparison with conventional approach without any ultrasound guidance.

DETAILED DESCRIPTION:
Peripheral venous catheter placement is one of the most common interventions in emergency medicine. When performed by conventional approach, the failure of the first attempt occurs up to 22 % and cannulation time exceed 2 minutes in up to 15 %. Ultrasound guidance of peripheral venous catheter (PVC) insertion may improve both. However, this approach has not been verified in the setting of pre-hospital emergency care so far.

ELIGIBILITY:
Inclusion Criteria:

* Awake patient indicated for peripheral venous catheter placement while treated by emergency medical service

Exclusion Criteria:

1. Coma
2. Age <18 years
3. Patient disagreement with the insertion of peripheral venous catheter
4. Disagreement of the patient with inclusion in a clinical trial
5. Contraindication of ultrasound examination of the venous system
6. Contraindication of the introduction of peripheral venous cannula on both upper limbs
7. Investigator's opinion that ultrasonic control cannulation would cause undue delay and a other procedure is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Frequency of the patients with successful the first cannulation attempt of peripheral venous catheter insertion | 60 minutes
  Frequency of the patients in which only one cannulation attempt was necessary

SECONDARY OUTCOMES:
Frequency of the patients with successful peripheral venous catheter insertion irrespective of the number of attempts | 60 minutes
  Frequency of the patients in which peripheral venous catheter was inserted, irrespective of the number of attempts
The number of attempts required for successful peripheral venous catheter insertion | 60 minutes
  The number of attempts required for successful peripheral venous catheter insertion
Time required to introduce peripheral venous catheter | 60 minutes
  Time required to introduce peripheral venous catheter

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Emergency Medical Service of Central Bohemian Region, Kladno, Czech republic
Locations (1):
- Emergency Medical Service of the Central Bohemian Region, Beroun, Central Bohemia, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Completely anonymous sharing of IPD
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 1.5.2018, two months
Access Criteria: investigator